CLINICAL TRIAL: NCT07388225
Title: The Effect of Preoperative Education on Recovery of Thoracic Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Eda Çiftçi Karan, Principal Investigator, Surgical Nursing, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THORACIC-EDU-RECOVERY-01
Record Dates: First submitted 2026-01-23; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer; Nursing Care; Patient Education; Thoracic Surgery
Keywords: Preoperative Education; Quality of recovery; Thoracic surgery; Pulmonary function test; Shoulder joint range of motion
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either an intervention group receiving structured preoperative education or a control group receiving routine care, and outcomes are assessed in parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: Structured Preoperative Education (Experimental): Participants assigned to this arm receive structured, nurse-led preoperative education in addition to routine hospital care prior to thoracic surgery.
  Interventions: Behavioral: Structured Preoperative Education
- Control Group: Routine Care (Active Comparator): Participants assigned to this arm receive standard preoperative and postoperative care routinely provided by the hospital.
  Interventions: Other: routine care

INTERVENTIONS:
Behavioral: Structured Preoperative Education — A structured, nurse-led preoperative education program delivered prior to thoracic surgery.
  Arms: Intervention Group: Structured Preoperative Education
Other: routine care — Standard care routinely provided by the hospital
  Arms: Control Group: Routine Care

SUMMARY:
Brief Summary

This randomized controlled study evaluated the effect of structured preoperative education on postoperative recovery outcomes in patients undergoing thoracic surgery for lung cancer. The study was conducted in a tertiary public hospital in Istanbul between June 2022 and December 2023 and included 100 adult patients who met the inclusion criteria. Participants were randomly assigned to an intervention group or a control group.

Patients in the intervention group received structured, nurse-led preoperative education supported by a standardized patient education booklet, while the control group received routine hospital care. Recovery outcomes were assessed using physiological parameters, pulmonary function tests, shoulder joint range of motion measurements, pain intensity scores, and the Quality of Recovery-40 (QoR-40) questionnaire during the early postoperative period.

The findings of this study aim to contribute evidence on the role of preoperative nursing education in improving functional recovery, reducing postoperative pain, and supporting respiratory function in patients undergoing thoracic surgery.

DETAILED DESCRIPTION:
Detailed Description

Thoracic surgery for lung cancer is associated with significant postoperative pain, reduced pulmonary function, limited shoulder mobility, and delayed functional recovery. These factors may negatively affect patient outcomes, prolong hospitalization, and increase the risk of postoperative complications. Preoperative education is considered a key nursing intervention that may enhance patients' physical and psychological preparedness for surgery and improve postoperative recovery.

This randomized controlled experimental study was conducted in the thoracic surgery units of a tertiary public hospital in Istanbul. A total of 100 patients scheduled for elective thoracic surgery due to lung cancer were enrolled and randomly assigned to either the intervention group (n=50) or the control group (n=50). Randomization was performed using a computer-generated randomization method.

Patients in the control group received standard preoperative and postoperative care routinely provided by the hospital. Patients in the intervention group received structured preoperative education delivered by a nurse, supported by a standardized patient education booklet. The education included information on the surgical procedure, breathing and coughing exercises, use of incentive spirometry, early ambulation, shoulder and upper extremity exercises, and pain management strategies.

Data were collected at three time points: preoperatively, on postoperative day 1, and on postoperative day 4. Outcome measures included pulmonary function tests (FEV1 and FVC), shoulder joint range of motion assessed by goniometry, pain intensity measured using the Visual Analog Scale (VAS), and recovery quality evaluated using the Quality of Recovery-40 (QoR-40) questionnaire. Vital signs and oxygen saturation levels were also recorded.

The primary objective of the study was to determine whether structured preoperative education improves postoperative recovery outcomes compared to routine care. Secondary objectives included evaluating the effects of education on pain levels, pulmonary function, shoulder mobility, and quality of recovery.

The results of this study are expected to provide evidence supporting the integration of structured preoperative nursing education into clinical care protocols for patients undergoing thoracic surgery, with the goal of improving functional recovery and patient-centered outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with lung cancer who are hospitalized for elective thoracic surgery
* Aged 18 years and older
* Able to read, write, and speak Turkish
* Able to understand the information provided and without any condition that interferes with verbal communication
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Patients scheduled for lung resection via thoracotomy
* Patients undergoing surgery under general anesthesia

Exclusion Criteria:

* Patients with chronic pain in the preoperative period who are using analgesic medications for pain management
* Patients receiving antineoplastic treatment
* Patients undergoing reoperation due to lung cancer
* Patients with an ECOG performance status greater than 2
* Patients diagnosed with metastatic lung cancer
* Patients with limited mobility in the preoperative period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative Recovery Quality | Postoperative day 1 and postoperative day 4
  Postoperative recovery quality assessed using the Quality of Recovery-40 (QoR-40) questionnaire. The total score ranges from 40 to 200, with higher scores indicating better recovery quality.

SECONDARY OUTCOMES:
Postoperative Pain Intensity | Preoperative period, postoperative day 1, and postoperative day 4
  Pain intensity assessed using the Visual Analog Scale (VAS), ranging from 0 to 10, where higher scores indicate worse pain.
Pulmonary Function | Preoperative period, postoperative day 1, and postoperative day 4
  Pulmonary function assessed using forced expiratory volume in one second (FEV1) and forced vital capacity (FVC), measured in liters.
Shoulder Joint Range of Motion | Preoperative period, postoperative day 1, and postoperative day 4
  Shoulder joint range of motion measured using a goniometer and expressed in degrees. Higher values indicate better functional outcome.
Postoperative Heart Rate | Preoperative period, postoperative day 1, and postoperative day 4
  Heart rate measured in beats per minute (bpm). Higher values indicate a worse outcome.
Postoperative Blood Pressure | Preoperative period, postoperative day 1, and postoperative day 4
  Systolic and diastolic blood pressure measured in millimeters of mercury (mmHg). Higher values indicate a worse outcome.
Postoperative Respiratory Rate | Preoperative period, postoperative day 1, and postoperative day 4
  Respiratory rate measured as breaths per minute. Higher values indicate a worse outcome.
Postoperative Oxygen Saturation | Preoperative period, postoperative day 1, and postoperative day 4
  Peripheral oxygen saturation measured by pulse oximetry and expressed as percentage (%). Higher values indicate a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, başakşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as this is a single-center academic thesis study and the informed consent and ethics approval do not include provisions for public data sharing.